CLINICAL TRIAL: NCT07221396
Title: A Single-Arm Study of LDART, a Social Support Intervention for Stimulant Use Disorder
Brief Title: Single-arm Study of LDART for Stimulant Use Disorder
Acronym: LDART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: College on Problems of Drug Dependence (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000040872; EarlyCareer Investigator grant (Other Grant/Funding Number: College on Problems of Drug Dependence)
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Stimulant Use Disorder; Cocaine Use Disorder; Methamphetamine Use Disorder
Keywords: social support; digital intervention; mutual-help groups; stimulant use disorder; addiction recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDART (Experimental): Participants will be given access to LDART for 28 days.
  Interventions: Behavioral: LDART

INTERVENTIONS:
Behavioral: LDART — Let's Do Addiction Recovery Together! (LDART) is a web-based intervention designed to be used for a few minutes each night to reduce problematic substance use. It has three active ingredients: 1) daily recovery goal setting and tracking, 2) motivational video, audio, and written messages from individuals in recovery, and 3) information on several community-based addiction recovery groups (e.g., support groups).

SUMMARY:
The goal of this study is to evaluate the feasibility, acceptability, and preliminary efficacy of a digital intervention called LDART in adults with stimulant use disorder.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Currently reside in Connecticut, USA
* Have a smartphone that can send and receive text messages and have internet access that can be access over the course of a month
* Substance (Stimulant) Use Symptom Checklist ≥2, indicating past-year stimulant use disorder
* Had high frequency of cocaine use (≥5 days) in the past 28 days
* Have some self-reported desire to cut down or quit stimulants

Exclusion criteria:

* Unable to provide informed consent, as assessed by the consent quiz
* Unable to speak, read, or write in English
* Vulnerable population status
* Unlikely to be able to complete study procedures in the next 2-3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From enrollment to the final assessment time point (Day 56)
  The percentage of eligible participants who are enrolled relative to the total number of eligible potential participants who completed the screening.
Accrual rate | From enrollment to the final assessment time point (Day 56)
  The rate of enrollment, defined as number of participants enrolled per month.
Retention rate | From enrollment to the final assessment time point (Day 56)
  The percentage of enrolled participants who complete all study-related procedures (i.e., all three assessments).
Intervention engagement | From beginning the intervention (Day 1) to the end of the intervention period (Day 28)
  Number of nights enrolled participants completed the activities on the LDART website, out of 28 nights.
Intervention acceptability | The second assessment time point (post-intervention, Day 28)
  Rating scores on the end-user version of the Mobile App Rating Scale (uMARS). Total score range 1-5 with higher scores indicating a better quality app.

SECONDARY OUTCOMES:
Change from baseline in stimulant use frequency | Baseline (Day 0), Post-intervention (Day 28), 1-month post-intervention (Day 56)
  Change in self-reported number of days when any stimulants were used in the past 28 days, as measured using the Timeline Follow-back.
Change from baseline in number of recovery groups engaged with | Baseline (Day 0), Post-intervention (Day 28), 1-month post-intervention (Day 56)
  Self-reported number of recovery groups engaged with in the past 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan McCurdy, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No